CLINICAL TRIAL: NCT00409136
Title: Physician Alerts to Prevent DVT and Pulmonary Embolism in Hospitalized Patients
Brief Title: Multi-Center Human Alert Trial to Prevent DVT and PE
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Samuel Z. Goldhaber, MD, Brigham and Women's Hospital
Other Study IDs: 2005-P-002527
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis; Cancer; Surgery
Keywords: Alert; Deep Vein Thrombosis; Pulmonary Embolism; Venous Thromboembolism; Prophylaxis; Anticoagulation
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Neoplasms; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Alert: Physicians alerted about their high risk patients who are not receiving any VTE prophylaxis.
  Interventions: Behavioral: Human Alert
- No Alert: Physicians not alerted about their high risk patients who are not receiving any VTE prophylaxis.
  Interventions: Behavioral: Human Alert

INTERVENTIONS:
Behavioral: Human Alert — An alert from study staff informing a physician that his/her patient is at high risk for DVT and/or PE, but is not receiving any prophylaxis.

SUMMARY:
To evaluate physician response to human alerts that inform the clinician that his/her patient may be eligible for thromboprophylaxis. Medical records are reviewed to evaluate prescribing decision and to evaluate rates of venous thromboembolism.

DETAILED DESCRIPTION:
Background Information and Rationale for the Study:

Venous thromboembolism (VTE) is often avoidable in hospitalized patients because proven prevention strategies have been established for patients at risk. North American and European prophylaxis guidelines have been widely disseminated. However, despite intensive educational efforts, VTE prevention remains underutilized.

At Brigham and Women's Hospital, we undertook a comprehensive program aimed at increasing the frequency of VTE prophylaxis in high risk patients. This novel strategy required: 1) devising a risk score that reliably and quickly identified patients at high risk of VTE, and 2) conducting a randomized controlled trial in which high risk patients without prophylaxis were randomized into an intervention or control group. The intervention group's physicians received a single alert explaining that the patient was at high risk, was not receiving prophylaxis, and urged that prophylaxis be selected from a template of available pharmacological and mechanical options. In contrast, the control group's physicians received no alert.

Each of 8 common risk factors was weighted according to a point scale. At least 4 score points were required to be deemed at "high risk" for VTE.

3 of the 8 risk factors were considered major and were assigned a score of 3 points each:

1. Cancer
2. Prior VTE
3. Hypercoagulability

One of the 8 risk factors, surgery, was considered intermediate and was assigned a score of 2.

4 of the 8 risk factors were considered minor and were assigned a score of 1 point each:

1. Advanced age (> 70 years of age)
2. Obesity (Body Mass Index > 29)
3. Bed rest
4. Hormone replacement therapy or oral contraceptives

There were 2,506 patients in the randomized controlled trial of a computer alert: 1255 in the intervention group and 1251 in the control group. The incidence of symptomatic VTE at 90 days was high: 8.2% in the control group. This high incidence validates the 8 risk factor and point score methodology.

The intervention group had an overall 41% reduction in VTE, without any increase in major bleeding. There was a 60% reduction in the incidence of symptomatic pulmonary embolism.

Identification of Patients at Risk for Venous Thromboembolism (VTE):

A VTE risk profile will be computed for each hospitalized patient using 8 common risk factors. Each risk factor is weighted according to a point score. To be included in this trial, the point score must equal or exceed 4 points.

Minor (Low) Risk Factors (1 POINT each):

* Advanced Age (>70 years of age)
* Obesity (BMI >29, or the presence of the word "obesity" in admission exam notes)
* Bed rest / Immobility (not related to surgery)
* Female Hormone Replacement Therapy or Oral Contraceptives

Intermediate Risk Factor (2 POINTS each):

· Major Surgery (> 60 minutes)

Major (High) Risk Factors (3 POINTS each):

* Cancer (active)
* Prior VTE
* Hypercoagulability

Increased VTE risk is defined as a cumulative VTE risk score 4, so that patients with at least 1 major risk factor (cancer, prior VTE, or hypercoagulability) plus at least 1 additional intermediate risk factor (major surgery or bed rest) or minor risk factor (advanced age, obesity, or hormone replacement therapy/oral contraceptives) become eligible. In the absence of a major risk factor, patients with 1 intermediate risk factor plus at least 2 minor risk factors become eligible.

Screening for Venous Thromboembolism Prophylaxis:

If the cumulative VTE risk score is ³4, orders are reviewed to detect ongoing mechanical or pharmacological prophylactic measures. Mechanical prophylactic measures include graduated compression stockings and intermittent pneumatic compression devices. Pharmacological prophylactic measures include unfractionated heparin, enoxaparin, dalteparin, fondaparinux, tinzaparin, and warfarin.

Randomization:

Randomization Envelopes containing the statement "ALERT" (Intervention) or "NO ALERT" (Control) will be provided by Harvard Clinical Research Institute (HCRI), to randomize patients who meet all inclusion criteria.

The intervention is informing the responsible physician that: 1) his or her patient is at high risk for VTE, 2) is not receiving prophylaxis, and 3) VTE prophylaxis is recommended. For control patients, VTE prevention guidelines are available, but no specific prompt is provided to use them.

Follow Up:

Ninety-day follow-up is performed in all study patients by medical record review and through contact with the subject's Primary Care Physician.

Data Collection and Study Endpoints:

The primary endpoint is clinically diagnosed DVT or PE at 90 days. Safety endpoints include total mortality and hemorrhagic events at 30 and 90 days, respectively. We define major bleeding as intracranial, intraocular, retroperitoneal, pericardial, or bleeding that requires surgical intervention or that resulted in a hemoglobin loss greater than 3 g/l.

DVT is diagnosed if there is loss of vein compressibility by ultrasound or a filling defect by CT scan or by conventional contrast venography. PE is diagnosed by a positive contrast chest CT scan, a high-probability ventilation perfusion scan, or conventional pulmonary angiogram.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Cumulative VTE risk score > 4
* Absence of pharmacologic or mechanical prophylaxis orders
* Patients from medical or surgical Services

Exclusion Criteria:

* VTE risk score <4
* Current active pharmacologic or mechanical prophylaxis order
* Patients from the Department of Neurology, Newborn Service, Rehab Units, and Neonatal Intensive Care Unit (NICU).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients that have a cumulative VTE risk score of 4 or more with no orders for prophylactic measures.
Sampling Method: Probability Sample
Enrollment: 2496 (Actual)
Dates: Start 2006-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Clinically diagnosed DVT and/or PE | 90 days

SECONDARY OUTCOMES:
Mortality | 30 and 90 days
Hemorrhagic events | 30 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Z. Goldhaber, MD, Principal Investigator — Brigham and Women's Hospital
Locations (26):
- United States (26):
  - AZ Pulmonary Specialists, Ltd, Scottsdale, Arizona
  - Long Beach VA Hospital, Long Beach, California
  - University of California - Irvine, Orange, California
  - University of California - Davis, Sacramento, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - William W. Backus Hospital, Norwich, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Hospital, Orlando, Florida
  - Emory-Crawford Long Hospital, Atlanta, Georgia
  - Franklin Square Hospital, Baltimore, Maryland
  - Washington County Hospital, Hagerstown, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - North Shore Medical Center, Salem, Massachusetts
  - Henry Ford Hospital K15, Detroit, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - University of Missouri, Columbia, Missouri
  - North Shore University Hospital, Great Neck, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson Hospital, Philadelphia, Pennsylvania
  - Washington Hospital, Washington, Pennsylvania
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - LDS Hospital, Salt Lake City, Utah
  - University of Utah Medical Center, Salt Lake City, Utah
  - United Hospital System, Kenosha, Wisconsin

REFERENCES:
- [Background] Goldhaber SZ, Turpie AG. Prevention of venous thromboembolism among hospitalized medical patients. Circulation. 2005 Jan 4;111(1):e1-3. doi: 10.1161/01.CIR.0000150393.51958.54. No abstract available. PMID 15630031
- [Background] Goldhaber SZ, Dunn K, MacDougall RC. New onset of venous thromboembolism among hospitalized patients at Brigham and Women's Hospital is caused more often by prophylaxis failure than by withholding treatment. Chest. 2000 Dec;118(6):1680-4. doi: 10.1378/chest.118.6.1680. PMID 11115458
- [Background] Goldhaber SZ, Tapson VF; DVT FREE Steering Committee. A prospective registry of 5,451 patients with ultrasound-confirmed deep vein thrombosis. Am J Cardiol. 2004 Jan 15;93(2):259-62. doi: 10.1016/j.amjcard.2003.09.057. PMID 14715365
- [Background] Kucher N, Koo S, Quiroz R, Cooper JM, Paterno MD, Soukonnikov B, Goldhaber SZ. Electronic alerts to prevent venous thromboembolism among hospitalized patients. N Engl J Med. 2005 Mar 10;352(10):969-77. doi: 10.1056/NEJMoa041533. PMID 15758007
- [Derived] Piazza G, Rosenbaum EJ, Pendergast W, Jacobson JO, Pendleton RC, McLaren GD, Elliott CG, Stevens SM, Patton WF, Dabbagh O, Paterno MD, Catapane E, Li Z, Goldhaber SZ. Physician alerts to prevent symptomatic venous thromboembolism in hospitalized patients. Circulation. 2009 Apr 28;119(16):2196-201. doi: 10.1161/CIRCULATIONAHA.108.841197. Epub 2009 Apr 13. PMID 19364975
- See also: North American Thrombosis Forum — http://www.natfonline.org/